CLINICAL TRIAL: NCT04738864
Title: The Effect of Behcet's Disease on Cerebrovascular Circulation
Brief Title: Neuro-ultrasound Assessment in Behcet's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Talaat, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17300548
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behcet's disease patient (Experimental): patient who presented with manifestation of behcet disease
  Interventions: Diagnostic Test: ultrasound
- Healthy people (Experimental): healthy control people
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — extracranial and intracranial ultrasound assessment

SUMMARY:
Assessment of structural changes that occur in large extracranial and intracranial arteries in patients with Behcet's disease

DETAILED DESCRIPTION:
Patients will be selected from Rheumatology and Rehabilitation inpatient and outpatient clinics in Assiute University Hospital Patients under 16 years old, patients with hyperlipidemia, hypertension, diabetes mellitus and all other risk factors affecting blood vessel intimal thickness will be excluded from the research.

All patients and control groups underwent a complete extracranial and intracranial ultrasound assessment by 2 experienced neurovascular sonographers .The ultrasound examination was done at the Neurovascular Ultrasound Laboratory in the Neurology department, Assiut University hospitals using a color-coded duplex ultrasound device Philips HD5 (Philips Medical Systems, Nederland B.V.) for the carotid and vertebral arteries and for the intracranial arteries.

Intimal medial thickness (IMT) of the common carotid artery (CCA), peak systolic velocities (PSVs) and end diastolic velocities (EDVs) were measured in the common, internal, and external carotid arteries (CCA, ICA, ECA) with L 3-12 MHz linear transducer probe and when stenosis was detected the velocities were measured at the maximally stenotic area.

The intracranial arteries were evaluated in all patients with transcranial color-coded duplexsonography (TCCS) with the use of a low-frequency (2- to 5-MHz) phased-array probe through the transtemporal acoustic bone window. The middle cerebral artery (MCA), intracranial segment of vertebral artery (V4)and basilar artery (BA) were examined. Peak systolic velocity (PSV) and flow direction (antegrade or reversed) used for the diagnosis of any intracranial atherosclerotic disease (ICAD).

The findings and the atherosclerotic changes in the extracranial and intracranial vessels were interpreted according to the internationally published data Data will be analyzed using the computer program SPSS

ELIGIBILITY:
Inclusion Criteria:

* patient more than 18 years old
* All patients fulfill the modified International Criteria for Behçet's Disease

Exclusion Criteria:

* Patients under 16 years old,
* patients with hyperlipidemia, hypertension, diabetes mellitus and all other risk factors affecting blood vessel intimal thickness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
CNS vascular involving | 6 mounth
  ultrasound of CNS vescle

CONTACTS AND LOCATIONS:
Overall Officials: Esraa A Talaat, Lecturer, Study Chair — Assiut University
Locations (1):
- Medicine, Asyut, Egypt